## Informativa e manifestazione del consenso al trattamento dei dati personali e di categorie particolari di dati personali ai sensi del Regolamento UE 2016/679

Titolo dello studio: METFORMIN CONTINUATION SAFETY IN DIABETIC PATIENTS UNDERGOING CORONARY ANGIOGRAPHY – studio NO-STOP

### Titolari del trattamento e relative finalità

Il Centro di sperimentazione IRCCS Istituto Clinico Humanitas - Humanitas Mirasole S.p.A., con sede legale in Rozzano (Milano), Via Alessandro Manzoni 56, (di seguito il "**Promotore dello studio**"), che ha commissionato lo studio che Le è stato descritto nel consenso informato al trattamento sanitario, ciascuno per gli ambiti di propria competenza e in accordo con la normativa in tema di tutela dei dati personali (Regolamento UE 2016/679 e Linee Guida per i trattamenti dei dati personali nell'ambito delle sperimentazioni cliniche dei medicinali del 24 luglio 2008), nonché in accordo nonché in accordo alle responsabilità previste dalle norme della buona pratica clinica (Decreto Legislativo 211/2003) e dalle norme in materia di studi clinici osservazionali (Circolare Ministeriale 6/2002), tratteranno i Suoi dati personali, in particolare la Sua storia clinica e le informazioni che verranno raccolte sottoponendoLa agli esami e agli accertamenti medici illustrati nello stesso consenso informato al trattamento sanitario. Altri dati relativi alla Sua origine e ai Suoi stili di vita verranno trattati solo ove indispensabili per la realizzazione dello studio o per fini di farmacovigilanza.

Non è previsto alcun trasferimento dei suoi dati personali al di fuori dell'Unione Europea. A tal fine, i dati indicati saranno raccolti e conservati presso il Centro di Sperimentazione.

Il trattamento dei dati personali relativi al Suo stato di salute ed alla Sua storia clinica è indispensabile per lo svolgimento dello studio, tale trattamento è basato sul Suo libero consenso: il rifiuto di prestarlo non Le consentirà di parteciparvi.

Se decide di non acconsentire al trattamento dei suoi dati personali, ciò non comporterà alcun pregiudizio sul tipo di cura o terapia che le è stata/verrà prescritta e somministrata.

## Modalità di elaborazione dei dati

I suoi dati saranno elaborati sia elettronicamente sia manualmente, saranno utilizzati per svolgere calcoli statistici. I risultati dello studio potranno essere pubblicati in pubblicazioni scientifiche, statistiche, convegni scientifici. In nessun caso i suoi dati potranno essere diffusi a tal fine se non in forma anonima.

La sua partecipazione allo Studio comporta che, in conformità alla normativa sulle sperimentazioni cliniche dei medicinali, il personale del Promotore dello studio, il Comitato Etico e Autorità sanitarie italiane e straniere possano essere informati circa i dati che la riguardano, compresi quelli presenti nella cartella clinica originaria, ma in modo tale da garantire la riservatezza sulla sua identità.

## Base Giuridica

La liceità del presente trattamento si basa sul consenso al trattamento dei propri dati personali di cui all'articolo 6, comma 1, lettera a) del Regolamento UE 2016/679 e sulla manifestazione del consenso

esplicito e informato da parte del soggetto interessato al trattamento di categorie particolari di dati personali, ai sensi dell'articolo 9 paragrafo 2 lettera a) del Regolamento UE 2016/679.

#### Natura dei dati trattati

Per quanto riguarda i suoi dati direttamente identificativi (ad es. nome, cognome) essi verranno trattati solo dal Centro di Sperimentazione. I dati inoltrati al promotore dello studio o ad altri enti indicati nel presente documento conterranno un codice al posto del Suo nome, per preservare la riservatezza della Sua identità: questi dati sono definiti "dati codificati".

Pertanto, il medico che La seguirà nello studio La identificherà con un codice: i dati che La riguardano raccolti nel corso dello studio, ad eccezione del Suo nominativo, saranno trasmessi al Promotore dello studio, registrati, elaborati e conservati unitamente a tale codice. Soltanto il medico e i soggetti autorizzati potranno collegare questo codice al Suo nominativo.

Tutti i dati presso di Lei raccolti verranno trattati con l'adozione di adeguate misure di sicurezza ex art. 32 ("Misure di Sicurezza) del Regolamento UE 679/2016.

## Tempi di conservazione dei dati

I suoi dati saranno conservati per un periodo massimo di 15 anni dalla conclusione della sperimentazione, ovvero dal momento in cui Lei decida di abbandonare lo studio, dopo di che saranno distrutti.

#### Esercizio dei diritti e dati di contatto del DPO

Lei ha diritto ad esercitare ognuno dei diritti previsti dal Regolamento Europeo 2016/679 a tutela dei soggetti interessati dal trattamento di dati personali, salvo le deroghe previste per i trattamenti per scopo di ricerca scientifica. In particolare:

- le è sempre riconosciuto il **Diritto di Accesso** ai sensi dell'Articolo 15 del Regolamento, ovvero il diritto di ottenere dal Titolare la conferma che sia o meno in corso un trattamento dei suoi dati personali e, in tal caso di ottenere, l'accesso ad una serie di informazioni sul trattamento in corso (come ad esempio: le finalità, le categorie di dati, i destinatari a cui sono comunicati e i suoi diritti);
- ha diritto di ottenere la **Rettifica dei dati personali** inesatti ai sensi dell'Articolo 16 del Regolamento;
- ha diritto di ottenere la **Cancellazione dei dati personali** che la riguardano nelle ipotesi previste dall'Articolo 17 del Regolamento, salvo che la cancellazione dei suoi dati non rischi di rendere impossibile o pregiudicare gravemente il conseguimento degli obiettivi di ricerca scientifica;
- ha diritto di ottenere la **Limitazione del trattamento** nei casi previsti dall'articolo 18 del Regolamento;
- ha il diritto di **opporsi al trattamento** nei casi previsti dall'Articolo 21 salvo che il trattamento sia necessario per l'esecuzione di un compito di interesse pubblico;
- ha il diritto di **revocare il suo consenso** in qualsiasi momento senza pregiudicare la liceità del trattamento basata sul consenso prestato prima della revoca,

Tali diritti e, in particolare il diritto alla cancellazione dei dati e il diritto di opporsi al trattamento, possono subire delle limitazioni qualora la cancellazione dei dati che la riguardano possano compromettere e pregiudicare il raggiungimento delle finalità illustrate.

In qualunque momento potrà esercitare i diritti di cui sopra scrivendo direttamente al Centro di Sperimentazione oppure al DPO del Centro al seguente indirizzo: Data Protection Officer dell'Istituto Clinico Humanitas - Via Manzoni 113, 20089 Rozzano (Milano) oppure all'indirizzo e-mail dataprotectionofficer@humanitas.it.

Inoltre, resta sempre salvo il suo Diritto di Reclamo all'Autorità Garante per la protezione dei dati personali.

Potrà interrompere in ogni momento e senza fornire alcuna giustificazione la Sua partecipazione allo studio. Non saranno inoltre raccolti ulteriori dati che La riguardano, ferma restando l'utilizzazione di quelli eventualmente già raccolti per determinare, senza alterarli, i risultati della ricerca.

## Modalità con cui potrà accedere alle informazioni contenute nel progetto di ricerca

In qualsiasi momento Lei potrà accedere alle informazioni contenute nel progetto di ricerca rivolgendosi al Centro di Sperimentazione all'indirizzo sopra indicato

# MODULO PER IL CONSENSO AL TRATTAMENTO DEI DATI PERSONALI E SANITARI

| Il/La sottoscritto/a |
|---|
| dichiara di aver letto e compreso l'informativa sul trattamento dei dati personali, inclusi dati relativi alla salute, che precede e in particolare di essere stato informato in merito a: |
| l'identità del Titolare del trattamento dei dati, |
| le modalità con le quali il trattamento avviene, |
| la base giuridica del trattamento, |
| la natura del conferimento dei dati, la natura dei dati trattati e le finalità del trattamento, |
| i tempi di conservazione dei Suoi dati |
| <ul> <li>i propri diritti, incluso il diritto di reclamo all'Autorità Garante,</li> <li>i dati di contatto del DPO</li> </ul> |
| □ ACCONSENTE □ NON ACCONSENTE |
| Ai sensi e per gli effetti dell'Articolo 6 paragrafo 1 lettera a) e ai sensi dell'Articolo 9 paragrafo 2 lettera a) del Regolamento Europeo 2016/679 al trattamento dei dati personali e dei dati sanitari secondo le modalità e nei limiti di cui alla presente Informativa. (1) |
| (Data) (Firma Del Soggetto Interessato) |

(1) Da sottoporre agli interessati unitamente al modulo di consenso informato che descrive le caratteristiche scientifiche dello studio, anche mediante integrazione dello stesso.